CLINICAL TRIAL: NCT01881360
Title: Comparison Between a Gluten-free Diet and a Hypocaloric Diet for the Treatment of Patients With Fibromyalgia and Celiac-type Symptoms
Brief Title: Efficacy of a Gluten-free Diet for the Treatment of Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Elena Pita Calandre, Responsible of the CTS-502 Investigation Team, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMS-GFD-013
Record Dates: First submitted 2013-06-17; First posted 2013-06-19 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; celiac-type symptoms; gluten-free diet; hypocaloric diet
MeSH Terms: conditions — Fibromyalgia | interventions — Diet, Gluten-Free

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gluten-free diet (Experimental)
  Interventions: Other: Gluten-free diet
- Hypocaloric diet (Active Comparator)
  Interventions: Other: Hypocaloric diet

INTERVENTIONS:
Other: Gluten-free diet — A diet that is free of the gluten component
  Arms: Gluten-free diet
Other: Hypocaloric diet — A standard hypocaloric diet with a daily 1500 caloric intake.
  Arms: Hypocaloric diet

SUMMARY:
Fibromyalgia patients frequently suffer from symptoms similar to those of adult celiac disease, raising the possibility that some fibromyalgia patients experience oligosymptomatic celiac disease or non-celiac gluten intolerance. The objective of this study is to compare the effect of a gluten-free diet with a hypocaloric diet in patients with fibromyalgia and celiac-type symptoms.

DETAILED DESCRIPTION:
Fibromyalgia, a chronic pain disorder, is characterized by generalized chronic musculoskeletal pain that is usually accompanied by several other clinical manifestations that contribute to a diminished quality of life, such as sleep disturbances, chronic fatigue, mood disorders, and cognitive difficulties. Many patients with fibromyalgia suffer from gastrointestinal and extra-intestinal symptoms that are similar to those experienced by adult celiac disease patients such as abdominal pain, dyspepsia, nausea, diarrhea, constipation, fatigue, pain and mood changes. This raises the possibility that some patients with fibromyalgia may also suffer from oligosymptomatic celiac disease or non-celiac gluten intolerance. On the other hand, the emerging evidence linking obesity with fibromyalgia and the high prevalence of overweight among fibromyalgia patients suggest a potential benefit for weight loss among these patients. Thus, the main objective of this study is to compare the efficacy of a gluten-free diet (GFD) with a hypocaloric diet (HCD) in patients with fibromyalgia that also experience celiac-type symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with fibromyalgia according to the 1990 American College of Rheumatology diagnostic criteria.
* Patients who successfully complete the screening process for sufficient celiac-type symptoms
* Negative transglutaminase antibodies serological testing.
* Signed informed consent to participate

Exclusion Criteria:

* Patients suffering from any disease that could prevent them from following any of the suggested diet protocols
* Current or previous history of substance abuse
* Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change, between baseline and endpoint, in the number of experienced celiac-type symptoms | 0, 4, 8, 12, 18 and 24 weeks

SECONDARY OUTCOMES:
Change, between baseline and endpoint, in the Body Mass Index | 0, 4, 8, 12, 18 and 24 weeks
Change, between baseline and endpoint, in the Revised Fibromyalgia Impact Questionnaire total score | 0, 4, 8, 12, 18 and 24 weeks
Change, between baseline and endpoint, in the Pittsburgh Sleep Quality Index | 0, 4, 8, 12, 18 and 24 weeks
Change, between baseline and endpoint, in the Brief Pain Inventory | 0, 4, 8, 12, 18 and 24 weeks
Change, between baseline and endpoint, in the Beck Depression Inventory | 0, 4, 8, 12, 18 and 24 weeks
Change, between baseline and endpoint, in the Short-form Health Survey | 0, 4, 8, 12, 18 and 24 weeks
Change, between baseline and endpoint, in the State-Trait Anxiety Inventory | 0, 4, 8, 12, 18, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena P. Calandre, M.D., Principal Investigator — Universidad de Granada
Locations (1):
- Instituto de Neurociencias "Federico Oloriz", Granada, Granada, Spain